CLINICAL TRIAL: NCT06381414
Title: Childhood Early Oral Aging Syndrome: Prevalence, Associated Etiological Factors, and Consequences on Vertical Dimension of Occlusion (VDO): A Cross-Sectional Study
Brief Title: Childhood Early Oral Aging Syndrome: Prevalence, Etiological Factors, and Consequences on Occlusion
Status: Recruiting | Type: Observational
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Other Study IDs: ChildhoodEarlyOralAging
Record Dates: First submitted 2024-04-17; First posted 2024-04-24 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Aging
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Observation — Identify the prevalence of early wear in primary dentition, using Childhood Early Oral Aging Syndrome (CEOAS) index.
  The CEOAS index involves scores of 0 to 3 for the assessment of tooth wear and dental management, whereas scores of I, II and III are used concomitantly in cases of the presence of enamel defects.

SUMMARY:
The Early Oral Aging Syndrome (EOAS) is a broad concept concerning changes in oral health caused by systemic diseases of different origins, which are related to the current lifestyle in the pediatric population. Enamel defects associated with intrinsic and extrinsic factors promote the acceleration of dental structure loss in an early manner, causing impairment of function, aesthetics, and quality of life. In this context, this study aims to identify the prevalence of early childhood tooth wear and its severity using the Early Childhood Oral Aging Syndrome (EOAS) index as a diagnostic and epidemiological survey instrument, considering current alterations found in the pediatric population and verifying possible factors associated with each severity level. Participants aged 3 to 6 years old, enrolled in the pediatric dentistry clinic of the University Nove de Julho, will be selected. Children with imperfect amelogenesis and dentinogenesis, genetic syndromes, and undergoing orthodontic treatment will be excluded from the research. A questionnaire on general health, sleep quality, nutrition, hygiene habits, and parafunctional habits will be administered. Subsequently, a clinical examination will be conducted using the new Early Childhood Oral Aging Syndrome (EOAS) index with scores ranging from 0 to 3 to assess dental wear and dental management, and scores I to III that should be used concomitantly in cases of enamel defects presence, in addition to measuring the Vertical Dimension of Occlusion (VDO). EOAS scores will be computed and statistically analyzed for deciduous dentition with a significance level of P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Children from three to six years of age with complete deciduous teeth;
* Children regularly enrolled for dental care at the Uninove pediatric dentistry clinic

Exclusion Criteria:

* Children with amelogenesis or dentinogenesis imperfecta
* Children undergoing orthodontic treatment
* Children with a genetic syndrome

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children regularly enrolled for dental care at the Uninove pediatric dentistry clinic
Sampling Method: Probability Sample
Enrollment: 183 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Assessment of Tooth Wear and Dental Management | Baseline
  CEOAS 0 - Absence of signs
  CEOAS 1 - Mild: Presence of clinical signs in reversible stages, without sensitivity. Such cases require follow-up.
  CEOAS 2 - Moderate: Presence of advanced signs with sensitivity and compromised function. Such cases require restorative treatment and management of the sensitivity.
  CEOAS 3 - Severe: Presence of severe signs with pulp involvement and the risk of the loss of the tooth. Such cases require more invasive and rehabilitative treatment.
Presence of Enamel Defects | Baseline
  CEOAS I- Presence of PMH - Demarcated opacities
  CEOAS II - Presence of PMH - Post-eruption fractures
  CEOAS III - Presence of fluorosis
Vertical Dimension of Occlusion | Baseline
  The VDO measurement will be carried out with the participant sitting, head aligned with the body and gaze fixed on a specific point. Measurements will be taken in centric occlusion and will be done with the aid of a digital caliper: The following distances will be measured with the aid of a digital caliper: 1° Distance from the corner of the lip to the corner of the eye; 2° Distance from the base of the nose to the chin.

CONTACTS AND LOCATIONS:
Locations (1):
- Nove de Julho University, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Spinola SG, Sobral APT, Mandetta ARH, Gimenez T, Goncalves MLL, Soares PV, Santos EM, Imparato JCP, Horliana ACRT, Mesquita-Ferrari RA, Motta LJ, Fernandes KPS, Bussadori SK. Childhood early oral ageing syndrome: prevalence and association with possible aetiological factors and consequences for the vertical dimension of occlusion: protocol for a cross-sectional study. BMJ Open. 2024 Dec 23;14(12):e090085. doi: 10.1136/bmjopen-2024-090085. PMID 39719276